CLINICAL TRIAL: NCT05583799
Title: The Efficacy and Adverse Effects of Niraparib in Ovarian Cancer: a Prospective Real-world Product Registration Study.
Brief Title: Efficacy and Adverse Effects of Niraparib in Ovarian Cancer.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2022LSK-354
Record Dates: First submitted 2022-09-26; First posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-09

CONDITIONS: Ovarian Cancer
Keywords: niraparib; efficacy and adverse effects; real word; prospective; product registration study
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — 10ml blood samples of enrolled patients are collected at baseline and study endpoints respectively (only for enrolled patients who agree to blood sampling) for exploratory biological marker research and exploratory pharmacogenetic analysis. All collected specimens will be kept in the first affiliated Hospital of Xi'an Jiaotong University.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ovarian cancer is the second fatal gynecological cancer. More than 70% of ovarian cancer patients are diagnosed as advanced. Niraparib was approved by the National Medical Products Administration on December 27, 2019. It can be used as a maintenance treatment for adult patients with platinum-sensitive recurrent epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer after platinum-containing chemotherapy has achieved complete or partial remission. On September 10, 2020, niraparib became a poly ADP-ribose polymerase inhibitor approved in China and globally, which can be used as a single agent for the maintenance treatment of first-line and recurrent ovarian cancer regardless of the patient's biomarker status. On December 28, 2020, niraparib has been included in the new version of the medical insurance catalog. At present, most studies based on niraparib are randomized controlled trials (RCTs). RCTs often have strict inclusion and exclusion criteria and they are implemented in a highly standardized environment. Its internal validity is high, but the research results may not be able to be extrapolated to practice. This study is a prospective real-world study. In this study, based on the modified Response Evaluation Criteria in Solid Tumors v.1.1 criteria, we evaluated the use of niraparib in patients with ovarian cancer, fallopian tube cancer, or primary peritoneal cancer in the progression-free survival, overall survival, and objective control rate, etc. The safety and tolerability of niraparib and the impact on the quality of life of patients are evaluated. 10ml blood samples of enrolled patients are collected at baseline and study endpoints respectively (only for enrolled patients who agree to blood sampling) for exploratory biological marker research and exploratory pharmacogenetic analysis. Finally, the results will as a supplement to the conclusions of randomized controlled trials to provide better guidance for patients.

DETAILED DESCRIPTION:
1. Research status at domestic and foreign

   Ovarian cancer is the second fatal gynecological cancer. More than 70% of ovarian cancer patients are diagnosed as advanced. Standard treatments include optimal reduction surgery and platinum/taxane chemotherapy. Epithelial ovarian cancer (EOC) is the most common histological type of ovarian cancer, up to 20% of high-grade serous ovarian cancer shows germline and/or somatic mutations in the BRCA1/BRCA2 gene. BRCA1 and BRCA2 are tumor suppressor genes that play a central role in repairing DNA double-strand breaks (DSB) through homologous recombination (HR). Due to their increased sensitivity to DNA damage reagents, they extend the survival period of BRCA1 and BRCA2 mutant EOCs, among which BRCA2 vectors have the best survival rate. Poly-ADP-ribose polymerase (PARP) 1 is a key ribozyme involved in single-strand break repair through the base excision repair pathway. In the absence of PARP activity, these lesions are considered to have transformed into DSB. Cells lacking HR, such as BRCA mutant cells, are extremely sensitive to PARP inhibition. This phenomenon called "synthetic lethality" has led people to study PAPP inhibitors used as therapeutic agents in BRCA1/BRCA2 carriers.

   Niraparib was approved by the National Medical Products Administration on December 27, 2019. It can be used as a maintenance treatment for adult patients with platinum-sensitive recurrent epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer after platinum-containing chemotherapy has achieved complete or partial remission. On September 10, 2020, niraparib became a PARP inhibitor approved in China and globally, which can be used as a single agent for the maintenance treatment of first-line and recurrent ovarian cancer regardless of the patient's biomarker status. On December 28, 2020, niraparib has been included in the new version of the medical insurance catalog. The results of the international phase III clinical trial (NOVA) of niraparib showed that niraparib can prolong the median progression-free survival of ovarian cancer patients regardless of whether the patients have germline BRCA mutations. Among patients with gBRCA mutations, the risk of disease progression was reduced by 73% and progression-free survival was 4-fold longer than in the placebo group (21 months vs. 5.5 months). In patients without the gBRCA mutation, the risk of disease progression was reduced by 55% and progression-free survival was more than 2-fold longer (9.3 months vs 3.9 months). The PRIMA clinical study showed that niraparib, as single-agent maintenance therapy, can significantly prolong the progression-free survival of first-line platinum-responsive ovarian cancer patients. The risk of disease progression and death was reduced by 38% across all treated patient populations. In BRCA-mutated, HRD-positive, and HRD-negative patients, niraparib reduced the risk of disease progression or death by 60%, 57%, and 32%, respectively. This study proves that niraparib becomes the first PARP inhibitor that can significantly improve the progression-free survival of patients regardless of biomarker status, which is expected to change the treatment of ovarian cancer in China. Recently, the first all-round, multicenter phase III clinical study in a Chinese population (NORA) showed that in patients with gBRCA mutations, median progression-free survival (PFS) was significantly longer with niraparib as second-line maintenance therapy, compared with placebo (not reached vs. 5.5 months, HR: 0.22) and those without gBRCA mutation at ESMO 2020(11.1 vs. 3.9 months, HR: 0.40). The QUADRA study shows that niraparib has a substantial survival benefit in women treated for ovarian cancer, especially in HRD-positive platinum-sensitive patients, including not only BRCA-mutated patients but also the BRCA wild-type population.

   The above-mentioned studies based on niraparib are mostly randomized controlled trials (RCTs). Because RCTs often have strict inclusion and exclusion criteria, they are carried out in a highly standardized environment, so that the research subjects have good homogeneity. The validity is high, but the research results may not be able to be extrapolated to practice. Therefore, it is necessary to evaluate the role of treatments for advanced diseases in the real environment. To provide better guidance for patients, real-world evidence is needed to make up for the lack of randomized controlled trials. At present, in real-world research, there are only retrospective studies on the use of niraparib in ovarian cancer at home and abroad, and the results are consistent with their corresponding RCTs. There is a lack of prospective real-world evidence with higher levels of evidence.
2. Study drugs

   The drug name is niraparib Tosylate capsules. This product is a 100mg capsule.
3. Research programs

   3.1 Overall design

   This study is a prospective real-world product registration study. It is an observational study. The main research content is to evaluate the efficacy and adverse reactions of PAPP inhibitors niraparib in patients with ovarian cancer, fallopian tube cancer, or primary peritoneal cancer. According to the inclusion and exclusion criteria, we collect various information about the target research participants, organize the data and perform statistical analysis under the guidance of epidemiologists and statistical experts. The curative effect is evaluated by indicators such as PFS, overall survival, and objective response rate. Moreover, we collect and analyze the adverse reactions of study participants after taking niraparib. 10ml blood samples of enrolled patients are collected at baseline and study endpoints respectively (only for enrolled patients who agree to blood sampling) for exploratory biological marker research and exploratory pharmacogenetic analysis.

   3.2 Sample size

   This research is an observational study. 222 study participants are expected to be included.

   3.3 Stratification factors

   This research can set up different plans according to the following different stratification factors and research purposes.1) Number of treatment lines: first-line maintenance, second-line maintenance, back-line treatment, excess indications. 2) BRCA1/2 mutation status: positive, negative. 3) Platinum sensitive status: platinum sensitive, platinum resistant. 4) carbohydrate antigen 125 (CA125) level, etc.

   3.4 Treatment plan

   This study is a non-interventional study that only collects data and does not interfere with clinical treatment. The medication is administered according to clinical instructions, guidelines, and local treatment routines.
4. Research process

   4.1 Subject informed

   Patients should sign an informed consent form before the start of the study. The researchers need to explain the contents of the informed consent to the subjects in detail. After the candidate has fully read and understood the informed consent, if she agrees to participate in the study, the subject should sign and date the informed consent. Researchers also need to sign and date the informed consent form.

   4.2 Interview on selection

   Within 7 days of the subjects' enrollment, the investigator collected baseline data, including general information; medical history diagnosis; past tumor treatment history; family history; whether it meets the admission criteria.

   4.3 Interview during treatment and the last interview
   * After the subjects are enrolled, the investigator will conduct a visit every 12 weeks. The data include: Efficacy evaluation: computed tomography/magnetic resonance imaging examination and tumor marker CA125 examination are required.
   * Safety evaluation: whether there are adverse events (AE).
   * At baseline, at the same time as the Response Evaluation Criteria In Solid Tumors assessment time (once every 12 weeks) until the objective radiation disease progression or the end of the study treatment interview, a functional assessment of cancer treatment-ovarian cancer questionnaire survey.
5. Safety evaluation

   5.1 Definition of Adverse Events

   AE refers to all the adverse medical events that occur after the subject receives the experimental drug. It can be manifested as symptoms and signs, diseases, or abnormal laboratory tests, but it may not be causally related to the experimental drug.

   5.2 Severity of adverse events

   During the study period, the severity of AEs will be classified according to Common Terminology Criteria for Adverse Events version 5.0, and AE of grade ≥3 will be collected.

   5.3 Relationship with study drug

   When judging the correlation between AEs and study drugs, the following factors should be considered: 1) It is definitely related; 2) It may be related; 3) Possibly irrelevant; 4) Definitely irrelevant; 5) Undecidable.

   5.4 Adverse event records

   All adverse events that occur from the subject's first use of niraparib to 4 weeks after the last dose, including observed by the investigator, obtained by inquiries, and spontaneously reported by the subject should be fully recorded.

   Researchers need to continue to follow up all AEs until the event is cured, returns to baseline, reaches a stable state, or no more information is available. The researcher needs to monitor and record the outcome of the AE in the subject's source file. After the study, there is no need to actively collect new AEs.
6. Drug management

   This study is a real-world study, and niraparib is a marketed drug, so niraparib needs to be purchased and used by patients according to the normal procedures in the hospital.
7. Data recording and monitoring

   7.1 Data logging

   This project uses table records. According to Good Clinical Practice requirements, in order to ensure patient privacy, patient names should not appear. All patients' names should be filled with name codes, and the codes should be abbreviated in Chinese names. The specific dosage and time of medication are unknown and should be filled in unknown rather than blank or missing items. The researcher should ensure that all data must be consistent with the "inpatient medical record".

   7.2 Data monitoring

   During the test process, the research unit will review the completed test case data, check whether the data is correct, complete, and standardized, and assess the traceability of all data.
8. Statistical analysis

   8.1 Definition of statistical analysis data sets

   The study includes cases that have received at least one trial drug and have a safety evaluation in the primary and secondary endpoint analysis. Those who have not used a trial drug or have no research data after being selected can be eliminated. Excluded cases should be kept for future reference and no statistical analysis should be performed.

   8.2 Statistical analysis methods

   The continuous variables in this study are described by median and interquartile ranges. Categorical variables are described by absolute value and the proportion of the total number of patients. Χ2 test is used for comparison between groups. The method of survival analysis is used to statistically process the follow-up data. Kaplan-Meier method is used to draw the survival curve of the follow-up subjects. The log-Rank test was used to evaluate the survival difference between each group. The Cox regression model was used to analyze the influencing factors of the survival time of each group of follow-up subjects. Candidate influencing factors with a significance level of 0.05 in the univariate analysis were selected for the multivariate analysis. For all analyses, the test level α=0.05, when p<0.05 is considered statistically significant. All analyses were performed using Statistical Product and Service Solutions software (version 22.0).
9. Quality control and quality assurance

All research processes should establish standardized operating procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary ovarian cancer, fallopian tube cancer, or peritoneal cancer confirmed by histology.
2. Patients who are taking niraparib.
3. Age greater than or equal to 18 years old.
4. Patients should voluntarily participate in the trial and provide signed informed consent.

Exclusion Criteria:

1.Patients who are not currently taking niraparib treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary ovarian cancer, fallopian tube cancer, or peritoneal cancer confirmed by histology
Sampling Method: Non-Probability Sample
Enrollment: 222 (Estimated)
Dates: Start 2022-10-15 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 24 months
  Progression-free survival is defined as the time from the first day of niraparib administration to disease progression (defined as objective radiological disease progression using modified Response Evaluation Criteria in Solid Tumors v.1.1 criteria or clinical progression) or death.
Incidence of Adverse Events | 24 months
  Adverse events classified according to Common Terminology Criteria for Adverse Events version 5.0.

SECONDARY OUTCOMES:
Overall survival | 60 months
  Overall survival is defined as from the first day of administration of niraparib to death of any cause or the patient's last follow-up.
Objective response rate | 24 months
  Objective Response Rate is defined as the percentage of patients with Complete Response or Partial Response, as assessed by Response Evaluation Criteria in Solid Tumors v.1.1 criteria using an independent review.
Health-related quality of life (HRQoL). | 24 months
  The functional assessment of cancer treatment-ovarian cancer (FACT-O) test result index (TOI) is used to assess the health-related quality of life of patients reported.

CONTACTS AND LOCATIONS:
Overall Officials: Qiling Li, Ph.D, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University